CLINICAL TRIAL: NCT02703181
Title: A Randomized, Placebo-controlled, Double-Blind (Sponsor Unblind), Repeat Dose, Ascending Cohort, Dose Escalation Phase I Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Epelsiban and Its Major Metabolite in Healthy Women Volunteers Following Administration of Repeat Dosing of Epelsiban
Brief Title: Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Epelsiban Administered in Repeat Doses in Healthy Women Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 201752
Record Dates: First submitted 2015-06-17; First posted 2016-03-09 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Embryo Transfer
Keywords: Safety; Dose Escalation; Repeat Dosing; Epelsiban; Pharmacokinetics; Healthy Women Volunteers; Tolerability; Oxytocin
MeSH Terms: interventions — epelsiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1(600 mg Epelsiban or placebo[every 8 hours]) (Experimental): Each subject will receive 200 mg of epelsiban administered TID (every 8 hours) (total daily dose of 600 mg) or a matching placebo administered every 8 hours.
  Interventions: Drug: Epelsiban (GSK557296); Drug: Placebo to match GSK557296

INTERVENTIONS:
Drug: Epelsiban (GSK557296) — White to off-white 0.270 inches x 0.700 inches oblong film coated tablet containing 25 mg or 100 mg epelsiban. To be swallowed whole with water, not to be chewed.
Drug: Placebo to match GSK557296 — White to off-white 0.270 inches x 0.700 inches oblong film coated Tablet containing placebo. To be swallowed whole with water, not to be chewed.

SUMMARY:
The current study is designed to assess the safety, tolerability and pharmacokinetics (PK) of additional repeat doses of epelsiban in healthy females, and will be the first dosing experience of repeat dosing at higher doses in women with this compound.

This study is a 14 day, randomized, placebo-controlled, double blind (sponsor unblind), repeat dose, ascending cohort, dose escalation study in healthy, female volunteers. Upon successful completion of the Screening period, a subject will be enrolled in the study. The study will be composed of three periods: Screening, Treatment and Follow-up. A subject's total time involved in the study will be approximately six weeks.

Cohorts will be conducted sequentially. Each subject will be enrolled in only one cohort. Ten subjects will be enrolled in each cohort and randomized to epelsiban (n=8) or placebo (n=2).

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 55 years of age inclusive, at the time of consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, review of medications previously used, physical examination, laboratory tests and electrocardiogram (ECG).
* Body mass index (BMI) within the range 18 - 35 kilogram per squared meter (kg/m^2) (inclusive)
* Not pregnant (as confirmed by a negative serum human chorionic gonadotropin [hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: Pre-menopausal females, postmenopausal, or women of reproductive potential who agree to follow one of the options listed in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential.

Exclusion Criteria:

* History of clinically significant abnormal transvaginal ultrasound
* Alanine aminotransferase (ALT) and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) > 450 milliseconds (msec)
* History of regular alcohol consumption within three months of dosing on Day 1 defined as: an average weekly intake of >7 drinks. One drink is equivalent to 12 gram (g) of alcohol: 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within three months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a known to inhibit or induce Cytochrome P450 3A4 [P450 CYP3A4]) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within three months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within three months
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2015-09-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time from time zero to infinite time (AUC[0 to infinity]) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose ante meridiem (AM), Pre Dose post meridiem (PM), Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Area under the concentration versus time from time zero to last time point with measurable concentration (AUC [0-t]) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Area under the concentration-time curve over the dosing interval (AUC [0-tau]) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Maximum observed concentration (Cmax) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Time of occurrence of Cmax (tmax) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Terminal phase half-life (t1/2) for epelsiban and GSK2395448 | Up to Day 15 (Day 1, 7 and 14)
  Blood samples were collected for Cohort 1 and 2 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, Pre- Dose PM2 (second PM dose [16h]), 0.5, 1, 2, 6, 8.5, 10, 14, 16.5, 17 and 24 hours post dose. Blood samples were collected for Cohort 3 on Days 1, 7, and 14 at Pre-dose AM, Pre Dose PM, 0.5, 1, 4, 6, 8, 12.5, 13, 16 and 24 hours post dose.
Safety as assessed by the number of subjects with adverse events (AE) and serious adverse events (SAE) | Up to Day 25
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of Subjects with clinically-significant changes in physical examination findings | Up to Day 25
  A complete physical examination will include, at a minimum, assessment of the cardiovascular (CV), respiratory, gastrointestinal and neurological systems. Weight will also be measured and recorded; height will only be measured and recorded at Screening.
Number of Subjects with clinically-significant changes in electrocardiograms (ECG) | Up to Day 15
  12-lead ECGs will be obtained after the subject has rested in the semi-supine position for at least 15 minutes. Triplicate 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals.
Blood pressure (BP) as a measure of safety and tolerability | Up to Day 15
  Triplicate readings of systolic and diastolic blood pressure will be obtained at each time point in semi-supine position after five minutes of rest.
Pulse rate measurements as a measure of safety and tolerability | Up to Day 15
  Triplicate readings of pulse rate will be obtained at each time point in semi-supine position after five minutes of rest.
Number of subjects with abnormal laboratory parameters | Up to Day 15
  Clinical laboratory assessments will include hematology, clinical chemistry and urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mahar KM, Enslin MB, Gress A, Amrine-Madsen H, Cooper M. Single- and Multiple-Day Dosing Studies to Investigate High-Dose Pharmacokinetics of Epelsiban and Its Metabolite, GSK2395448, in Healthy Female Volunteers. Clin Pharmacol Drug Dev. 2018 Jan;7(1):33-43. doi: 10.1002/cpdd.363. Epub 2017 May 26. PMID 28556598
- See also: Results for study 201752 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201752?search=study&b'search_terms=201752'#rs